CLINICAL TRIAL: NCT04467255
Title: Muscular Fatigue Evaluation in Patients With Diabetic Neuropathy by Means of Multichannel Surface Electromyography After a Rehabilitative Training: Aerobic Versus Endurance Training.
Brief Title: Surface Electromyography Study of Fatigue in Diabetic Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CE 2185
Record Dates: First submitted 2020-06-23; First posted 2020-07-10 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Neuropathy; Diabetes Mellitus
Keywords: sEMG, diabetic neuropathy, fatigue, training
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Neuropathies; Fatigue

STUDY DESIGN:
Intervention Model Description: Participants are assigned to two groups in parallel for the duration of the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group a (Active Comparator): aerobic training
  Interventions: Other: Rehabilitative training
- group b (Active Comparator): endurance training
  Interventions: Other: Rehabilitative training

INTERVENTIONS:
Other: Rehabilitative training — 4 weeks aerobic treadmill training compared to endurance training with elastic thera band

SUMMARY:
Fatigue in diabetic neuropathy compromises patients' physical activity and poses questions on how to plan correct rehabilitation training. Conclusive interpretation of muscular mechanisms of fatigue in diabetic neuropathy has not yet been achieved. Among the various instrumental evaluations for fatigue, multichannel surface electromyography (sEMG) is a recognized tool that permits the study of myoelectric manifestations of fatigue. Aim of the study is to assess if differences in myoelectric manifestations of fatigue between patients affected by diabetic neuropathy exist after an aerobic or endurance training.

DETAILED DESCRIPTION:
The instrumental session consisted of the registration of sEMG signals during electrically stimulated and voluntary contractions according to a consolidated standardized protocol. The investigated muscle is the Anterior Tibial.

Each subjects sat comfortably on a chair with his/her ankle flexed at 90° degree and knee extended; the leg was fixed at 90 degrees, in the isometric brace fixed on a plane (MISO1, LISiN Bioengineering Centre, Turin Polytechnic, Italy Torque was measured with a modular brace incorporating two independent torque transducers (model TR11, CCT Transducers, Torino, Italy).

The signal from the two torque meters were amplified, summed and displayed by means of a visual feedback system, which provided the subject with information regarding the torque level produced. Torque signal were stored to be analysed later.

The sEMG signal of the right Anterior Tibial was investigated with a flexible adhesive linear array of 16 electrodes (silver bars 10 mm long, 1 mm diameter, 10 mm apart) in single differential (SD) configuration. The optimal position and orientation of the array was determined at moderate contraction levels by visual inspection of the signal. It provided clear motor unit action potentials with similar propagation in the two directions from the neuromuscular junction to the tendons.

The reference electrode was positioned on the patient's leg. The skin was cleaned by slightly abrading it with abrasive gel before positioning the array.

Since sEMG variables are affected by muscle temperature, the skin temperature was monitored with an electronic thermometer throughout the whole examination and was kept between 31.5 C° and 32.5 C° 30.

The protocol consisted in three evaluations: one stimulated contraction and two voluntary contractions, according to a standardized protocol.

The stimulated contraction was executed through a button stimulation electrode (size: 10 mm) positioned on the motor point using a monopolar configuration, a frequency of 25 Hz for a duration of 30 seconds and a supramaximal stimulation. The motor point was selected as the position of the stimulated electrode on the skin where the M-wave showed the maximum amplitude for a specified stimulation intensity; the supramaximal stimulation level was defined as the current intensity above which there was no significant increase of the amplitude of the M-wave or the maximum level tolerated by the subjects.

A rest period of 10 minutes after stimulation was observed in order to avoid cumulative fatigue phenomenon.

The subject then performed two test-contractions by dorsiflexion of the foot against the resistance given by the braces, in order to get acquainted with the procedure and to verify the correct posture and position of the array.

The subject was subsequently asked to produce three maximal voluntary contractions (MVC) lasting 3 seconds each with a rest period of 2 minutes in-between. The reference MVC, expressed in Nm, was established as the maximum of the three measurements. The last MVC measurement was followed by a 10-minute rest period.

The subject then produced two voluntary contractions each lasting 30 seconds: one contraction at 30% MVC and one at 60% MVC with a 5-minute rest in between. A visual biofeedback was used to help the subject maintaining the requested contraction level; furthermore, the subjects were verbally encouraged to obtain the best outcome during their performance.

The EMG signals were filtered with a 10-500 Hz bandwidth filter, amplified (EMG 16-16 channel amplifiers LISiN Bioengineering Centre Turin Polytechnic). They were sampled at 2048 Hz during voluntary contractions and 1024 Hz during electrically elicited contractions. Signals were digitised by a 16 bit A/D converter (DAQCARD-6024E National Instruments, Austin, Texas, USA) and stored on the disk of a personal computer.

Signal processing was performed using MATLAB. EMG variables of interest were: mean normalized frequency (MNF), average rectified value (ARV) and muscle fibre conduction velocity (CV). Spectral (i.e. MNF), amplitude (i.e. ARV) and CV variables were computed with numerical algorithms described in previous papers.

CV was estimated from the consecutive double differential signals showing the best signal propagation; MNF and ARV were estimated from the single differential channel in the middle of the channels used for CV estimation. Epoch length for EMG variable estimation was 0.5 seconds without overlapping.

A linear regression was used to fit all the scatter graphs of the EMG variables with time. The rate of change was defined as the slope of the regression line. The normalized rate of change for all variables was defined as the ratio between the slope and the intercept (initial value of sEMG variables) expressed as percentage. Physiological myoelectric manifestations of muscle fatigue consist in reduction of MNF and CV and increase of ARV.

ELIGIBILITY:
Inclusion Criteria:

* Michigan Neuropathy Screening instrument higher or equal to 7
* Stable clinical conditions

Exclusion Criteria:

* Other neurological conditions or diseases
* Skin lesions
* Recent lower limb fractures or lower limb surgical intervention

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-05-22 (Actual); Primary Completion 2024-07-16 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Six-minute walk test | 4 weeks
  The score of the test is the distance a patient walks in 6 minutes measured in meters.

SECONDARY OUTCOMES:
Modified Borg Scale | 4 weeks
  Is is commonly used to assess fatigue during a training expressed with Dyspnea. This is a0 to 10 rated scale. High score corresponds to worse outcome.
Functional Independence Measure | 4 weeks
  The functional Independence measure is an 18-item measurement tool that explores an individual's physical, psychological and social function. The tool is used to assess a patient's level of disability. Range total score 18-126. High score corresponds to better outcome.
Surface multichannel electromyographic variables. | 4 weeks
  In research setting muscle electric properties were analyzed during contractions employing multichannel surface electromyograpy. Among the variables describing muscle activity, we examine conduction velocity. The conduction velocity of the muscle was estimated from the difference in arrival time of the motor unit potential at electrodes separeted by 15 mm. The motor unit conduction velocity for anterior tibial, analyzed in this study, ranged from 2.6 to 5.3 m/s (mean 3.7 m/s) (Arendt-Nielsen SA and L. J Physiol (1987), 391, pp 561-571).

CONTACTS AND LOCATIONS:
Locations (1):
- Ics Maugeri, Montescano, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Callaghan BC, Cheng HT, Stables CL, Smith AL, Feldman EL. Diabetic neuropathy: clinical manifestations and current treatments. Lancet Neurol. 2012 Jun;11(6):521-34. doi: 10.1016/S1474-4422(12)70065-0. Epub 2012 May 16. PMID 22608666
- [Background] Chipkin SR, Klugh SA, Chasan-Taber L. Exercise and diabetes. Cardiol Clin. 2001 Aug;19(3):489-505. doi: 10.1016/s0733-8651(05)70231-9. PMID 11570119
- [Background] Fritschi C, Quinn L. Fatigue in patients with diabetes: a review. J Psychosom Res. 2010 Jul;69(1):33-41. doi: 10.1016/j.jpsychores.2010.01.021. Epub 2010 Mar 23. PMID 20630261
- [Background] Watanabe K, Gazzoni M, Holobar A, Miyamoto T, Fukuda K, Merletti R, Moritani T. Motor unit firing pattern of vastus lateralis muscle in type 2 diabetes mellitus patients. Muscle Nerve. 2013 Nov;48(5):806-13. doi: 10.1002/mus.23828. Epub 2013 Aug 30. PMID 23447092